CLINICAL TRIAL: NCT04456491
Title: The Clinical Value of the Nitric Oxide System Components in Asthma and Chronic Obstructive Pulmonary Disease
Brief Title: The Clinical Value of the Nitric Oxide System Components in Asthma and COPD
Acronym: ASCONO
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Ryazan State Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: ASCONO
Record Dates: First submitted 2020-06-29; First posted 2020-07-02 (Actual); Last update posted 2023-07-21 (Actual); Status verified 2023-07

CONDITIONS: Asthma; COPD
Keywords: nitric oxide, arginine, arginase
MeSH Terms: conditions — Asthma; Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — venous blood sample
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Asthma: Patients with Asthma
- COPD: Patients with COPD
- Control group: Healthy volunteers

SUMMARY:
It is planned to conduct a study of nitric oxide metabolites (nitrates and nitrites), L-arginine, arginase-1, and asymmetric dimethylarginine in patients with bronchial asthma and chronic obstructive pulmonary disease, followed by observation to assess the prognosis of the disease.

DETAILED DESCRIPTION:
Chronic obstructive pulmonary disease and bronchial asthma have a leading position among respiratory diseases. A significant contribution to the clinical picture and long-term prognosis is made by exacerbations of COPD, which makes it relevant to search for methods for their prediction and prevention. According to the global initiative on bronchial asthma (GINA), bronchial asthma is characterized by high heterogeneity and the existence of many phenotypes and endotypes, which makes it relevant to use personalized medicine methods in patient management and, in particularly, the search for new biomarkers of asthma. Currently, in clinical practice, some biomarkers of obstructive lung diseases are widely used. Among them there are the level of eosinophils in the blood and sputum, the level of immunoglobulin E and the exhaled fraction of nitric oxide (FeNO). Obstructive lung diseases are characterized by persistent inflammation in the airways, which is accompanied by the manifestation of elements of systemic inflammation and endothelial dysfunction, which is associated with an altered release of vasoactive mediators, one of them is nitric oxide (NO). NO is a powerful vasodilator that is synthesized from L-arginine using the enzyme NO synthase (NOS). The NO molecule has small lifetime from 3 to 30 s, that's why the search for biomarkers with a more stable lifetime is relevant. Some of them it's nitric oxide metabolites, such as nitrates (NO3-), nitrites (NO2-), S-nitrosothiols, 3-nitrotyrosine. Nitrates and nitrites, which are metabolites of nitric oxide, may be of interest as one of the promising biochemical markers reflecting NO metabolism in the human body. Earlier in our study, the relationship between the plasma level of nitric oxide metabolites and the severity of bronchial asthma was shown, which may be a prerequisite for further study of the components of the nitric oxide system as potential biomarkers of bronchial obstructive diseases.

A promising direction in the search for biomarkers related to the nitric oxide system is the study of L-arginine, which acts as a substrate in the reaction of NO formation. The bioavailability of L-arginine for NO synthases determines the activity of formation of nitric oxide in the respiratory tract, as evidenced by the effect of inhaled L-arginine on the level of exhaled fraction of nitric oxide. Earlier, in a US study, 26 patients with bronchial asthma showed a significant decrease in plasma L-arginine levels compared with healthy volunteers, and laboratory animal models showed that a decrease in L-arginine levels leads to airway hyperreactivity. Currently, a number of pilot clinical interventional studies have been carried out in which the administration of L-arginine improved the manifestations of bronchial asthma in some patients, but did not change the frequency of exacerbations in the total sample of patients. This indicates the possible existence of an endotype of bronchial asthma associated with impaired functioning of the nitric oxide system, and makes it promising to study the level of L-arginine in the blood as a potential biomarker of obstructive lung diseases.

In addition to studying nitric oxide metabolites, substances that affect the formation of NO should be considered as potential biomarkers of the disease. One such substance is arginase, under the influence of which L-arginine is converted into L-ornithine and urea. In humans, two isoenzymes of arginase, arginase 1 and arginase 2, have been identified, which differ in cellular location and tissue distribution. Both arginase enzymes are expressed in the airways and can be found in endothelial and epithelial cells, fibroblasts, macrophages, and smooth muscle cells of the respiratory tract. Further metabolism of L-ornithine leads to the formation of polyamines and L-proline, which are involved in cell proliferation and differentiation, as well as in the production of collagen. Scientists have shown that increased arginase activity in the airways contributes to airway obstruction and hyperreactivity by decreasing the availability substrate for NOS. As a result, the production of NO decreases and superoxides form, which react with NO to form peroxynitrite, thereby increasing airway contractility and inflammation. In addition, increased airway arginase activity leads to an increase in L-ornithine production, which potentially contributes to airway remodeling due to stimulation of cell proliferation and collagen formation.

The metabolism of L-arginine depends not only on arginase, but also on the methyltransferase enzyme, which methylates L-arginine residues, which undergo proteolysis with the formation of asymmetric and symmetric dimethylarginine (ADMA and SDMA). These amino acids inhibit NOS activity, since ADMA is a competitive inhibitor of the enzyme, while SDMA is a competitor to L-arginine transport. Serum ADMA and SDMA, as well as L-arginine concentrations increase with COPD and increase further with the development of exacerbation. It is important to note that the concentration of ADMA in blood serum is probably an independent risk factor for long-term mortality from all causes in obstructive lung diseases and is associated with increased airway resistance. In recent years, several studies have been conducted examining the association of ADMA with obstructive lung diseases. Earlier the association of ADMA with the development of obstructive lung diseases, airway resistance and indicators of the function of external respiration in patients with obstructive lung diseases was shown.

Thus, there are prerequisites for studying the components of the nitric oxide system, such as metabolites of nitric oxide, L-arginine, arginase, and asymmetric dimethylarginine, as a biomarker of obstructive lung diseases. Based on this, it is planned to study of nitric oxide metabolites (nitrates and nitrites), L-arginine, arginase-1, and asymmetric dimethylarginine in patients with bronchial asthma and chronic obstructive pulmonary disease, followed by observation to assess the prognosis of the disease.

The study is aimed at studying the clinical value of the nitric oxide synthesis modulators (L-arginine, arginase-1 and asymmetric dimethylarginine) in patients with bronchial asthma and chronic obstructive pulmonary disease, as well as assessing their effect on the prognosis and the course of diseases .

The study objectives is

1. To assess the levels of modulators of the synthesis of nitric oxide (L-arginine, arginase-1 and asymmetric dimethylarginine) in the blood of patients with asthma and chronic obstructive pulmonary disease and their relationship with the clinical course of the disease.
2. To evaluate the clinical value of the ratio of the levels of modulators of the synthesis of nitric oxide (L-arginine, arginase-1 and asymmetric dimethylarginine) and the level of metabolites of nitric oxide (nitrates and nitrites) in patients with bronchial asthma and chronic obstructive pulmonary disease.
3. To assess the possibility of using the determination of the levels of modulators of nitric oxide synthesis to predict the course of obstructive lung diseases and prevent the development of exacerbations of bronchial asthma and chronic obstructive pulmonary disease.
4. To assess the possibility of developing personalized treatment regimens for obstructive lung diseases, based on the assesment of the levels of modulators of the synthesis of nitric oxide (L-arginine, arginase-1 and asymmetric dimethylarginine) in the blood of patients with asthma and chronic obstructive pulmonary disease.

It is planned to conduct a prospective case-control study in the three study groups. To all patients will be performed: general clinical examination; Test of Adherence to Inhalers; clinical and biochemical analysis of the blood; spirometry; assesment of the level of nitric oxide metabolites in serum using the photocolorimetric method in Griss reaction; assesment of the level of L-arginine, arginase-1 and asymmetric dimethylarginine in serum by enzyme immunoassay using the laboratory kit Immundiagnostik (Germany). At the second phase of the study, lasting 2 years, the prognostic capabilities of assesment the levels of modulators of nitric oxide synthesis will be evaluated using a combined endpoint, included increase in level of basis therapy, exacerbation, hospitalisation and mors associated with Asthma and COPD.

ELIGIBILITY:
Inclusion Criteria:

* men and women aged between 18 and 70 years
* a diagnosis of asthma or chronic obstructive pulmonary disease according to actual GINA and GOLD guidelines

Exclusion Criteria:

* decompensated pathology of the cardiovascular system;
* history of liver dysfunction accompanied by an increase in ALT, AST or total bilirubin more than 3 times higher than the upper limit of normal;
* history of severe renal impairment, accompanied by a decrease in glomerular filtration rate below 60 ml/min (according to CKD-EPI);
* abuse on psychoactive substances and / or alcohol.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Asthma and COPD patients from Ryazan region which admitted in clinics of the Ryazan State Medical University
Sampling Method: Probability Sample
Enrollment: 240 (Estimated)
Dates: Start 2021-09-01 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Combined outcome - clinical worsening | 2 years
  Combined outcome including increase in level of basis therapy, exacerbation, hospitalisation and mors associated with Asthma and COPD

SECONDARY OUTCOMES:
NO-metabolites | At initial visit
  Serum level of total nitric oxide metabolites (nitrites and nitrates summary)
L-arginine | At initial visit
  Serum level of L-arginine
Arginase-1 | At initial visit
  Serum level of arginase-1
ADMA | At initial visit
  Serum level of asymmetric dimethylarginine

CONTACTS AND LOCATIONS:
Overall Officials: Anton Shakhanov, MD, Cand.Sci. (Med.), Principal Investigator — Ryazan State Medical University
Locations (1):
- Department of Therapy, Ryazan, Ryazanskaya Obl., Russia

IPD SHARING:
Plan to Share IPD: No